CLINICAL TRIAL: NCT01478022
Title: Open, Randomized, 3 Period Cross-over Design, in Healthy Volunteers to Compare the Pharmacokinetics Profiles of 3 Treatments: ISO 20, IBU 200 and IBU Plus ISO Combinations (200 + 20) Administered Per os as Single Doses
Brief Title: To Compare the Pharmacokinetics Profiles of ISO 20, IBU 200 and IBU Plus ISO Combinations 200 + 20
Acronym: ISOFEN1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parent Project, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISOFEN1
Record Dates: First submitted 2011-11-14; First posted 2011-11-23 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: DMD; Duchenne; Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Isosorbide Dinitrate; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Isosorbide Dinitrate 20 mg (Active Comparator): Isosorbide Dinitrate 10 mg b.i.d
  Interventions: Drug: Isosorbide Dinitrate
- Ibuprofen 200 mg (Active Comparator): Ibuprofen 200 mg daily, capsule
  Interventions: Drug: Ibuprofen
- Isosorbide dinitrate and Ibuprofen (Experimental): Isosorbide dinitrate 20 mg daily and Ibuprofen 200 mg daily
  Interventions: Other: Ibuprofen and Isosorbide Dinitrate combination

INTERVENTIONS:
Drug: Isosorbide Dinitrate — Isosorbide Dinitrate 10 mgx2, daily, capsules
  Other Names: Diniket 10 mg
  Arms: Isosorbide Dinitrate 20 mg
Drug: Ibuprofen — Ibuprofen 200 mg daily, capsules
  Other Names: Antalgil 200 mg
  Arms: Ibuprofen 200 mg
Other: Ibuprofen and Isosorbide Dinitrate combination — Ibuprofen 200 mg and Isosorbide Dinitrate 20 mg combination daily dose
  Other Names: Antalgil 200 mg and Diniket 10 mg
  Arms: Isosorbide dinitrate and Ibuprofen

SUMMARY:
This study will evaluate the pharmacokinetics plasma profile of 3 treatments: ISO 20, IBU 200 and IBU and ISO combinations (200 +20) given in single dose.

This study is being conducted to support the submission for new indication in treatment of the combinations of Isosorbide Dinitrate and Ibuprofen as a treatment for Duchenne muscular dystrophy.

DETAILED DESCRIPTION:
This trial is designed to define drug interactions following the combined administration of Isosorbide Dinitrate, a NO donor, and ibuprofen, NSAID, a through pharmacokinetics approach.

Both ibuprofen and Isosorbide Dinitrate were licensed worldwide. Ibuprofen is approved for use in adults and children; Isosorbide is approved for use in adults. Ibuprofen is currently used in pediatric patients as a first line anti-inflammatory and antipyretic agent. Consensus exists that among NSAIDs ibuprofen is the one endowed with less adverse effects (see note 66 of the Italian Drug Agency AIFA and MEA). No specific studies concerning safety and tolerability of ISDN in pediatric patients have been reported.

ELIGIBILITY:
Inclusion Criteria:

* Healthy free-living
* Males between the age of 18 and 27
* Normal ECG
* Body Mass Index of 19.0-29.0 (Kg/m2)
* Subject healthy in the opinion of the Investigator
* Signed informed consent after verbal and written information

Exclusion Criteria:

* Clinically significant underlying systemic illness that may preclude the subject's ability to complete the trial
* Any Gastrointestinal conditions which, in the opinion of the Investigator, may interfere with the absorption of the drug or render the subjects unable to take oral medication (gastric ulcer, peptic ulcer, stomach acid, frequent diarrhea, gastrointestinal surgery)
* History of the following cardiac diseases SBP <120 mmHG or DBP < 80 mmHg
* Platelet count < 100000/mm3
* History of recurrent headache
* History of ongoing or clinically relevant glaucoma
* History of alcohol, drug or medication abuse within the past 2 years
* Treatment with norepinephrine, acetylcholine and histamine
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* Participation in another study phase 1 with any investigational product within 6 months of screening

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: AUC 0-12 | At period I, II and III with 7 days intervals between periods
  Area under the time-concentration curve (AUC 0-12) of IBU and ISO given concomitantly compared to AUCs of ISO alone and IBU alone. Time points: = at pre dose, 30, 60, 90, 120, 150, 180, 210, 240 min and 5, 6, 8, 10 and 12 hrs post dose

SECONDARY OUTCOMES:
C max | At period I, II and III with 7 days intervals between periods
  C max of IBU and ISO given concomitantly compared to AUCs of ISO alone and IBU alone. Time points: = at pre dose, 30, 60, 90, 120, 150, 180, 210, 240 min and 5, 6, 8, 10 and 12 hrs post dose
T max | At period I, II and III with 7 days intervals beteween periods
  T max of IBU and ISO given concomitantly compared to AUCs of ISO alone and IBU alone. Time points: = at pre dose, 30, 60, 90, 120, 150, 180, 210, 240 min and 5, 6, 8, 10 and 12 hrs post dose
Adverse Events | 9 days
  Adverse Events registration At visit 2, visit 3 and visit 4
Vital signs | 9 days
  Pulse rate and blood pressure (Diastolic and Systolic) measurements in sitting position at pre-dose, and 1 and 3 hours after study drug intake. Complete physical examination At visit 2, visit 3 and visit 4

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Clementi, Principal Investigator — Luigi Sacco Hospital - Phase I Department - Via G. B. Grassi 74 20157 Milano
Locations (1):
- Clinical Phase 1 Unit - Luigi Sacco Hospital, Milan, Italy